CLINICAL TRIAL: NCT03988998
Title: radioFrequency Ablation With or Without RadioTherapy for Small HEpatocellulaR Carcinoma: a Randomized Control Trial
Brief Title: Radiofrequency Ablation Plus Radiotherapy for Small Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Professor, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FARTHER
Record Dates: First submitted 2019-06-13; First posted 2019-06-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Radiofrequency Ablation with or without Radiotherapy
Who Masked: Outcomes Assessor
Masking Description: Outcomes (recurrence or death) Assessor is blind about the interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency ablation with radiotherapy (Experimental): Patients in this arm will receive liver radiotherapy around the primary tumor margin within one month after radiofrequency ablation for hepatocellular carcinoma.
  Interventions: Drug: Radiofrequency ablation with radiotherapy
- Radiofrequency ablation alone (Active Comparator): Patients in this arm will only receive radiofrequency ablation for hepatocellular carcinoma.
  Interventions: Drug: Radiofrequency ablation alone

INTERVENTIONS:
Drug: Radiofrequency ablation with radiotherapy — Radiofrequency ablation with radiotherapy
  Arms: Radiofrequency ablation with radiotherapy
Drug: Radiofrequency ablation alone — Radiofrequency ablation without radiotherapy
  Arms: Radiofrequency ablation alone

SUMMARY:
Radiofrequency ablation (RFA) and hepatic resection are main treatments for early stage hepatocellular carcinoma. Many randomized controlled trials found these two treatments have similar short term overall survival. However, hepatic resection is associated with higher long-term overall survival. These results reveal that tumor recurrence rate after RFA is higher than that after hepatic resection. And minimal residual tumor may exist after RFA. Radiotherapy after RFA may be effective to prevent early tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnoses of hepatocellular carcinoma based on EASL.
2. Tumors, either single, >2 and < 5 cm in size or no more than 3 for size < 3 cm.
3. Patients must have a performance status of ECOG score < 2.
4. Patients must have adequate liver reservation and adequate hemogram.

   * Pugh-Child's Score < 7.
   * The serum total bilirubin level are < 2 mg/dl.
   * The prothrombin times are < 3 sec above normal control.
   * The platelet are > 75 x 109/L.
5. Patient must have serum creatinine < 1.5 mg/dl
6. Cardiac function with NYHA classification < Grade II
7. HBsAg (+) .
8. Signed informed consent.

Exclusion Criteria:

1. HCCs with radiological evidence of macrovascular invasion or extrehepatic metastasis are not eligible.
2. Patients with other systemic diseases which required concurrent usage of glucoticosteroid or immunosuppressant agent(s) are not eligible.
3. Patients with advanced second primary malignancy are not eligible.
4. Patients with pregnancy or breast-feeding are not eligible.
5. Patients with severe cardiopulmonary diseases are not eligible.
6. Patients with clinically significant psychiatric disorder are not eligible.
7. Patients who had antineoplastic chemotherapeutic or immuno-therapeutic drugs or corticosteroids within 6 weeks of commencing the protocol are not eligible.
8. Patients who had prior antitumor therapy for HCC are not eligible.
9. Anti-HCV positive patients are not eligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-10 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
the 2-years recurrence rate | 2 year
  Two year recurrence rate between the two groups will be compared.

SECONDARY OUTCOMES:
the 2-years recurrence-free survival | 2 year
  Two year recurrence-free survival between the two groups will be compared.
the 2-years overall survival. | 2 year
  Two year overall survival between the two groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Tang Wei-Zhong, PhD, Study Chair — Guangxi Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wahl DR, Stenmark MH, Tao Y, Pollom EL, Caoili EM, Lawrence TS, Schipper MJ, Feng M. Outcomes After Stereotactic Body Radiotherapy or Radiofrequency Ablation for Hepatocellular Carcinoma. J Clin Oncol. 2016 Feb 10;34(5):452-9. doi: 10.1200/JCO.2015.61.4925. Epub 2015 Nov 30. PMID 26628466
- [Background] Seo YS, Kim MS, Yoo HJ, Jang WI, Paik EK, Han CJ, Lee BH. Radiofrequency ablation versus stereotactic body radiotherapy for small hepatocellular carcinoma: a Markov model-based analysis. Cancer Med. 2016 Nov;5(11):3094-3101. doi: 10.1002/cam4.893. Epub 2016 Oct 5. PMID 27709795
- [Background] Hara K, Takeda A, Tsurugai Y, Saigusa Y, Sanuki N, Eriguchi T, Maeda S, Tanaka K, Numata K. Radiotherapy for Hepatocellular Carcinoma Results in Comparable Survival to Radiofrequency Ablation: A Propensity Score Analysis. Hepatology. 2019 Jun;69(6):2533-2545. doi: 10.1002/hep.30591. Epub 2019 May 2. PMID 30805950
- [Background] Kim N, Kim HJ, Won JY, Kim DY, Han KH, Jung I, Seong J. Retrospective analysis of stereotactic body radiation therapy efficacy over radiofrequency ablation for hepatocellular carcinoma. Radiother Oncol. 2019 Feb;131:81-87. doi: 10.1016/j.radonc.2018.12.013. Epub 2018 Dec 31. PMID 30773192